CLINICAL TRIAL: NCT01925963
Title: Development of Normative Datasets for Assessments Planned for Use in Patients With Mild Traumatic Brain Injury (NORMAL)
Brief Title: Normative Datasets for Assessments Planned for Mild Traumatic Brain Injury (NORMAL)
Acronym: NORMAL
Status: Completed | Type: Observational
Sponsor: Lindell Weaver (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); The Emmes Company, LLC (Industry); Intermountain Health Care, Inc. (Other); Evans Army Community Hospital (Other)
Responsible Party: Sponsor-Investigator, Lindell Weaver, Study Director, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Other Study IDs: S-11-16
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Focus: Healthy Adults Without Brain Injury
Keywords: Normal; Traumatic brain injury; Neuroimaging; Hyperbaric oxygen; Neurobehavioral symptom inventory
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma will be collected and frozen for future analyses. Future work may examine DNA, chronic neuro-response biomarkers, plasma- and leukocyte-based markers of TBI using a number of modern molecular techniques to examine the expression profiles of genes, proteins, and other macromolecules and to correlate these profiles to clinical outcomes, and genotypes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal cohort: Normal, healthy adults without history of brain injury

SUMMARY:
The purpose of the research study is to collect information about brain function and structure among active duty military personnel or civilians who are healthy. Researchers want to develop a database from normal volunteers that will be used in comparison with a similar database from active duty military with post-concussive syndrome (PCS) from a mild traumatic brain injury. Findings from this study may be used to design larger studies that will evaluate whether hyperbaric oxygen treatments actually improve PCS.

Participants in this study will undergo numerous tests to assess physical, mental, and intellectual health and how they might change over time. Participants will wear heart and activity monitors, undergo brain imaging, provide blood and urine for laboratory testing, and have vision, hearing, balance, and muscle function tests. They will also complete a number of questionnaires and interviews. This battery of tests will be repeated twice more over the course of 6 months.

DETAILED DESCRIPTION:
The primary purpose of this study will develop a database from normal healthy participants for the same outcomes used in a program of studies of hyperbaric oxygen (HBO2) vs. sham control in participants with persistent post-concussive symptoms. This study will characterize the distribution of responses and change in responses over time for each of the outcomes and will examine associations between measures within a given normal participant and across participant characteristics such as age and gender. It will evaluate the test-retest reliability of a series of assessments anticipated for use in the primary, secondary, and exploratory outcomes of this program of studies.

A secondary purpose of this study is to compare normative values to results from randomized exploratory studies of HBO2 vs. sham control in participants with persistent post-concussive symptoms. Also, investigators will examine relationships between outcome measures from normal participants (with respect to clinical equivalence, participant burden, and risk) and compare to associations observed in other studies.

In this study, normal, healthy, non-brain injured civilians and military participants (active or inactive) will undergo a battery of outcome assessments at defined test intervals to replicate the assessment battery used in a program of studies investigating the safety of HBO2 in patients with post-concussive symptoms following mild traumatic brain injury (TBI).

The planned comprehensive assessments will obtain robust neuropsychological, physiological, and neuroimaging data. Other evaluations will include laboratory testing and evaluations of the auditory, vestibular, and visual systems. Neuroimaging (magnetic resonance imaging and computed tomography angiography) will be assessed in participants at baseline and 6 months. Neurological function and electroencephalography (EEG) will be assessed at baseline only. All other in-person outcome measures will be assessed in participants at baseline, at 13 weeks, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Active duty or civilian in the Colorado Springs area.
* Men 18-65 years old and women 18-35 years old at the time of enrollment.
* Able to speak and read English, as primary language.
* Agrees to, and appears able to participate in all outcome assessments.
* Agrees to provide blood samples for laboratory tests and specimen banking.
* Demonstrates the ability to offer informed consent and signs the study informed consent document.
* No known brain imaging abnormalities.
* Known history of full term non-complicated birth.
* Estimated glomerular filtration rate (eGFR) >90.

Exclusion Criteria:

* Prisoners.
* Pregnant Women.
* Minors.
* Civilian participants with planned leave conflicting with study visits or relocation within 6 months of study enrollment, and unwilling or unable to return for follow up.
* Active duty participants with planned leave or deployment conflicting with assessment intervals.
* Any lifetime history of brain injury.
* Diagnosis of, or a persistent history of, or symptoms of a neurological disorder (e.g., tinnitus, vertigo, chronic fatigue, numbness, tingling, chronic migraine, fibromyalgia, multiple sclerosis).
* Active therapy for affective disorders, behavioral disorders, or psychological disorders.
* Diagnosis of diabetes mellitus
* Current complaints of brain injury symptoms such as cognitive or affective problems.
* Diagnosis of recurrent migraine or cluster headaches that are under medical management.
* Headaches that occur more than two times per week.
* Recurrent dizziness that requires medical management.
* Dizziness more than two times per week.
* History of theater or war zone activity that placed the participant within a combat zone environment.
* Diagnosis of PTSD or sub-clinical post-traumatic symptoms.
* Known neuroimaging abnormalities.
* Use of daily prescription drugs that could impact a normal outcome (e.g., beta blockers, antidepressants), with the following exceptions:
* Participants who are 45 or more years old may be taking statins or ACE inhibitors.
* Oral or injectable contraceptives are permitted
* Participants <45 years old who are taking any daily prescriptions (exception - oral or injectable contraceptives)
* Known atrial septal defect.
* History of hydrocephalus/microcephaly/macrocephaly.
* History of developmental delay or learning disorder as a child.
* Women who are breastfeeding.
* Women of childbearing potential who do not agree to practice an acceptable form of birth control during the study period.
* Allergy to iodine-based contrast dye (exclusion criteria for neuroimaging assessment measures).
* Those who are unable to participate fully in outcome assessments unless enrollment is reviewed and approved (in writing) by the Study Director.
* Binocular vision not correctable to 20/50.
* Deafness in both ears defined as 90 decibel hearing loss or greater through speech frequencies.
* Anxiety or claustrophobia precluding participation in neuroimaging or vestibular procedures.
* History of therapeutic ionizing radiation to the head.
* Foreign material in head that would interfere with brain imaging.
* Foreign material within the individual that poses risk from MRI.
* History of illicit drug use, except remote, non-habitual use of marijuana.
* History in the last year, of alcohol abuse.
* Current positive urine test for an illicit substance(s).
* Active or prior malignancy except basal cell carcinoma within the last 5 years.
* Unable to abstain from caffeine or tobacco products for at least a 2-hour interval.
* Concurrent enrollment in any other research trial.
* Unable or unwilling to cease participation in sports or activities in which head injury is likely (e.g., mixed martial arts, boxing) during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal, healthy, non-brain injured civilians and military participants (active or inactive)
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

PRIMARY OUTCOMES:
Change in neuropsychological test scores across time | Baseline and 13 weeks

SECONDARY OUTCOMES:
Change in neuropsychological test scores across time | Baseline and 6 months
Change in cerebral blood flow by computed tomography angiography | Baseline and 6 months
Change in brain anatomical structures by quantitative magnetic resonance imaging | Baseline and 6 months
Change in brain activation by functional magnetic resonance imaging | Baseline and 6 months
Change in visual refractive error | Baseline and 13 weeks
Change in visual refractive error | Baseline and 6 months
Change in sleep quality total score by Pittsburgh Sleep Quality Index | Baseline and 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Price, MD, Principal Investigator — Evans Army Community Hospital
Locations (2):
- United States (2):
  - Outcomes Assessment Center, Colorado Springs, Colorado
  - Evans Army Community Hospital, Colorado Springs, Colorado

REFERENCES:
- [Background] Weaver LK, Cifu D, Hart B, Wolf G, Miller S. Hyperbaric oxygen for post-concussion syndrome: design of Department of Defense clinical trials. Undersea Hyperb Med. 2012 Jul-Aug;39(4):807-14. PMID 22908837
- [Derived] Wetzel PA, Lindblad AS, Mulatya C, Kannan MA, Villmar Z, Gitchel GT, Weaver LK. Eye tracker outcomes in a randomized trial of 40 sessions of hyperbaric oxygen or sham in participants with persistent post concussive symptoms. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):299-311. PMID 31394600
- [Derived] Meehan A, Lewandowski A, Deru K, Hebert D, Weaver LK. Reference ranges and stability of auditory and vestibular measures in a comprehensive assessment battery for traumatic brain injury. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):227-241. PMID 31394594
- [Derived] Weaver LK, Wilson SH, Lindblad AS, Churchill S, Deru K, Price R, Williams CS, Orrison WW, Patel JB, Walker JM, Meehan A, Mirow S; NORMAL Study Team. Comprehensive Evaluation of Healthy Volunteers Using Multi-Modality Brain Injury Assessments: An Exploratory, Observational Study. Front Neurol. 2018 Dec 17;9:1030. doi: 10.3389/fneur.2018.01030. eCollection 2018. PMID 30631299
- [Derived] Walker JM, Mulatya C, Hebert D, Wilson SH, Lindblad AS, Weaver LK. Sleep assessment in a randomized trial of hyperbaric oxygen in U.S. service members with post concussive mild traumatic brain injury compared to normal controls. Sleep Med. 2018 Nov;51:66-79. doi: 10.1016/j.sleep.2018.06.006. Epub 2018 Jun 30. PMID 30099354
- [Derived] Wetzel PA, Lindblad AS, Raizada H, James N, Mulatya C, Kannan MA, Villamar Z, Gitchel GT, Weaver LK. Eye Tracking Results in Postconcussive Syndrome Versus Normative Participants. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):4011-4019. doi: 10.1167/iovs.18-23815. PMID 30098189